CLINICAL TRIAL: NCT02251002
Title: Frontoparietal Priority Maps as Biomarkers for MTBI
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1408M53005
Record Dates: First submitted 2014-09-22; First posted 2014-09-26 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: TBI (Traumatic Brain Injury); Ocular Motility Disorders
MeSH Terms: conditions — Brain Injuries, Traumatic; Ocular Motility Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: no history of TBI or neurologic disorder
- mTBI: documented past mild to moderate TBI

SUMMARY:
The purpose of this study is to determine whether there is a quantitative relationship between brain processes seen by a MRI and visual deficits caused by mild to moderate traumatic brain injuries (mTBI).

DETAILED DESCRIPTION:
Participants with mTBI, as well as healthy control participants, will be invited to participate in up to two study visits. Both visits will occur at the University of Minnesota's Center for Magnetic Resonance Research (CMRR). The first study visit will entail (1) interviews to determine the presence of (and, if present, the severity of) oculomotor difficulties such as convergence insufficiency, and (2) behavioral measures (e.g., visually track a moving dot) to assess skill at allocating spatial attention. For participants who have not before participated in an MRI study at the CMRR, a 15-minute scan to acquire research-quality anatomical images of the brain will be acquired at the end of the first visit. A subset of the approximately 88 participants who participate in Visit 1 will be invited to participate in Visit 2. Visit 2 will be dominated by a 90-minute scanning session in the 7 Tesla scanner, during which participants will perform a 10-minute spatial attention task and a 10-minute eye movement task, and high-resolution diffusion tensor imaging data will be acquired while participants enjoy the movie of their choice in the scanner.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected to normal visual acuity
* No previously documented mTBI (target: 16 out of 88 participants invited for Visit 1)
* Previously documented mTBI (target: 72 out of 88 participants invited for Visit 1)
* Vision impairment (target: 48 out of 88 participants invited for Visit 1; expected to be comorbid with mTBI, but non-TBI participants with oculomotor impairments will not be excluded)

Exclusion Criteria:

* Current use of neuroactive drugs or medications
* Presence of neurological disorders (other than mTBI and mild PTSD)
* Contraindications for MRI (metal in the body, claustrophobia, diabetes or other diseases or drugs that affect thermoregulation)
* Inability to comply with behavioral task instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with mTBI who have previously participated in MRI studies; preference will be given to individuals with visual complaints such as blurred or double vision or headaches while reading. Participants with no history of TBI and no visual complaints will also be recruited into a control group.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
oculomotor performance | study enrollment / baseline
  Oculomotor performance will be measured with behavioral questionnaires, eye-charts, and computerized eye-tracking while subjects perform saccades and smooth pursuit motions.

SECONDARY OUTCOMES:
frontoparietal priority maps | baseline
  Functional MRI data will be collected at 7 Tesla while subjects perform spatial attention and eye movement tasks.
white matter integrity | baseline
  Diffusion tensor imaging data will be acquired at 7 Tesla and analyzed in a priori regions of interest adjacent to frontal and parietal functional regions of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A Olman, PhD, Principal Investigator — University of Minnesota